CLINICAL TRIAL: NCT02326428
Title: An Open, Prospective, Blinded Evaluation, International, Multicentre, Controlled Study of Safety and Efficacy of Thrombectomy and Standard Stroke Care in Clinical Routine Treatment of Acute Occlusive Stroke Compared to Standard Stroke Care Only
Brief Title: SITS (Safe Implementation of Treatments in Stroke) Open Artery by Thrombectomy in Acute Occlusive Stroke Study
Acronym: SITS Open
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other); Medtronic - MITG (Industry); Stryker Nordic (Industry); Phenox GmbH (Industry)
Responsible Party: Principal Investigator, Nils Wahlgren, MD, PhD, FESO, Professor of Neurology, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SITS Open
Record Dates: First submitted 2014-05-21; First posted 2014-12-29 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Cerebrovascular Accident; Brain ischemia; Intravenous thrombolysis; Stroke thrombectomy; Stent-retriever
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia | interventions — Thrombectomy; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thrombectomy (Experimental): Thrombectomy arm consists of patients undergoing thrombectomy according to accepted critera in the judgement of investigator. Patients may be included even if they are not treated with intravenous thrombolysis because of contraindication or other reasons.
  Interventions: Device: Stent retriever endovascular device for thrombectomy; Drug: Intravenous thrombolysis by alteplase (Actilyse) (optional)
- Control (Active Comparator): Control arm patients are treated with standard stroke care including IVT but do not receive Thrombectomy. Control arm consists of patients fulfilling criteria for thrombectomy according to accepted critera in the judgement of investigator. Patients may be included even if they are not treated with intravenous thrombolysis because of contraindication or other reason.
  Interventions: Drug: Intravenous thrombolysis by alteplase (Actilyse) (optional)

INTERVENTIONS:
Device: Stent retriever endovascular device for thrombectomy — Thrombectomy by selected stent retrievers (TREVO, Solitaire, pREset, in special cases all stent retrievers) as additional therapy in major artery occlusion in patients fulfilling criteria for and receiving intravenous thrombolysis
  Other Names: Mechanical thrombectomy in ischemic stroke
  Arms: Thrombectomy
Drug: Intravenous thrombolysis by alteplase (Actilyse) (optional) — Stroke thrombolysis with Alteplase (Boeringer-Ingelheim, ATC-code B01AD02; a fibrinolytic drug) according to conventional guidelines (0.9 mg/kg, not exceeding 90 mg, given intravenously)
  Other Names: Stroke thrombolysis

SUMMARY:
Ischemic stroke, i.e. irreversible damage of a part of the patient's brain, is caused by the formation of blood clot in the major vessel which gives blood supply to a certain part of the brain. At early time, within the first 4,5 hours, the conventional treatment is to try to dissolve this blood clot with a medication ("thrombolytic drug") which is administered to the blood through the needle in the vein. If the clot still remains there, additional treatment is possible - going directly to the clot via artery and taking it out with a special device. Patients may be included even if they are not treated with intravenous thrombolysis because of contraindication or other reasons. The purpose of the present study is to evaluate the benefit and safety efficacy of thrombectomy and standard stroke care in clinical routine treatment of acute occlusive stroke compared to standard stroke care only.

ELIGIBILITY:
Inclusion criteria:

* Patients with acute stroke after exclusion of intracranial haemorrhage on CT/MRI scan.
* Confirmed diagnosis on CTA of persisting occlusion of the terminal Internal Carotid Artery (Car-T), proximal Middle Cerebral Artery (MCA, M1), proximal part of the insular segment of MCA (M2), proximal part of the anterior cerebral artery (A1), Basilar Artery (BA) or proximal part of the posterior cerebral artery (P1), consistent with the clinical symptoms. For inclusion in the study, CTA must not be performed later than 15 minutes after IVT start if given. For patients not treated with IVT, CTA should preferably be performed within 15 minutes of completion of the non-contrast CT but must be performed within 6 hours after stroke onset.
* Eligible patients for IVT are treated according to clinical guidelines (Attachment 1), and IVT, if given, initiated within 4.5 h.
* Initiation of thrombectomy is recommended within 6 hours after stroke onset but must be performed within to 8 hours if thrombectomy would still be of benefit for the patient as judged by the investigator.
* Baseline NIHSS Score at initiation of IVT is recommended between 7 and 25 for anterior circulation stroke and ≥7 without upper limit for posterior circulation stroke (baseline NIHSS score should be assessed by an NIHSS-certified physician), but patients may also be included beyond these scores if thrombectomy would still be of benefit for the patient as judged by the investigator.
* Age ≥18years.
* Anticipated life expectancy of at least 6 months.
* Patient or legal representative is competent to make a decision and has provided informed consent with regard to participation in the study, retrieval and storage of data and follow up procedures.
* Initiation of endovascular procedure (DSA/TBY, defined as start with groin puncture) within 2 hours from the start of IVT, or after CTA if IVT is not given (for TBY arm patients).

Exclusion criteria:

* Known significant pre-stroke disability (mRS ≥2).
* Extended early ischemic changes for basilar artery occlusion, according to the judgment of treating physician based on routine clinical practice of the hospital; if technical possibility exists, early irreversible ischemic changes may be confirmed by pc-ASPECTS score < 8 on CTASI (2) or extensive DWI lesion on pre-treatment MRI.
* Known pregnancy.
* Participation in any other investigational drug or device study, currently or in the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Categorical shift in modified Rankin Scale score at 3 months | 90 (range 76-104) days from stroke onset
  Categorical shift towards better stroke outcome as reflected by lower, i.e. better, Rankin Scale scores over the range of the scale in active compared to control group.

SECONDARY OUTCOMES:
Functional independence at 3 months after stroke onset | 90 (76-104) days after stroke onset
  Proportion of patients with functional independence (modified Rankin Scale, mRS, score 0-2) at 3 months after stroke onset
Excellent recovery at 3 months | 90 (76-104) days after stroke onset
  Proportion of patients with excellent outcome (mRS score 0-1) at 3 months
Length of in-hospital stay | 90 (76-104) days after stroke onset
  Days to discharge from in-hospital ward to home/secondary care for survivors in thrombectomy vs. control
Home time stay | 90 (76-104) days after stroke onset
  Number of days the patient stayed at home or at relative's stay within the first 3 months after stroke onset, in thrombectomy vs. control
Recurrent stroke within 3 months | 90 (76-104) days after stroke onset
Recanalisation of the occluded artery for thrombectomy treated population | 6h
  Recanalisation of the occluded artery for thrombectomy treated population, defined as at least TICI 2b flow in the treated territory after procedure
Time to revascularisation | 6h
  Time from stroke onset to revascularisation to any TICI (Thrombolysis in Cerebral Infarction) grade (2b-3 by core lab evaluation) for the actively treated population
Recanalisation of the occluded artery at 24h computerized tomography angiography /contrast-enhanced magnetic resonance angiography | 22-36h
  Defined as AOL 2-3
Proportion of patients with recanalisation before thrombectomy | 6h
  Defined as AOL 2-3
Reduction of infarct size | 22-36h
  Reduction in infarct size (thrombectomy vs. control) at 22-36 hours
Neurological and functional improvement in relation to thrombus length | 90 (76-104) days
  Neurological improvement (difference in National Institute of Health Stroke Scale from baseline to 12h, to 24h and to 7D after initiation of intravenous thrombolysis, or discharge if earlier), and functional outcome at 3 months in relation to recanalisation status and thrombus length (mm)
All-cause mortality at 3 months | 90 (76-104) days
Neurological death within 7 days post treatment | 7 days
Distal embolism/reocclusion demonstrated by follow-up computerized tomography angiography /contrast-enhanced magnetic resonance angiography | 22-36h
  Distal embolism/reocclusion will be evaluated by DSA immediately following the endovascular intervention and at the 22-36 hour follow up CT and CTA scans. The proportion of patients with recanalisation of the target occlusion and distal enbolism/reocclusion will be calculated.
Embolism into new territories (ENT) | 22-36h

OTHER OUTCOMES:
Symptomatic intracerebral haemorrhage (SICH) according to SITS-MOST definition | 22-36 h
  • Symptomatic intracerebral haemorrhage (SICH) according to SITS-MOST definition: local or remote parenchymal haemorrhage type 2 on the 22- to 36-hour post-treatment imaging scan, combined with a neurological deterioration of ≥4 points compared with baseline NIHSS or the lowest NIHSS value or death between baseline and 24 hours.
Symptomatic intracerebral haemorrhage (SICH) according to modified SITS-MOST definition | 22-36h
  • Symptomatic intracranial haemorrhage (SICH) according to modified SITS-MOST definition; in addition to usual SITS-MOST criteria blood may be anywhere in the intracranial space (including in the intraventricular, intraparenchymal and/or subarachnoid space).
Symptomatic intracerebral haemorrhage (SICH) according to modified ECASS III definition | 22-36h
  • Symptomatic intracranial haemorrhage (SICH) defined as an NIHSS decline of ≥4 points compared with baseline NIHSS or the lowest NIHSS value or death between baseline and 7 days, associated with any haemorrhage judged by core lab evaluation to be responsible for the decline. Blood may be anywhere in the intracranial space including in the intraventricular, intraparenchymal and/or subarachnoid space (modified ECASS III definition).
Number of adverse effects of thrombectomy | up to 90 (76-104) days
  Any adverse reactions related to thrombectomy procedure including patients for whom the initiating angiography revealed recanalisation by IVT only

CONTACTS AND LOCATIONS:
Overall Officials: Nils Wahlgren, Professor, Study Chair — Karolinska Institutet; Olav Jansen, Professor, Study Chair — University Hospital of Schleswig-Holstein; Staffan Holmin, M.D., Ph.D., Principal Investigator — Karolinska University Hospital, Karolinska Institutet; Kennedy Lees, M.D., FRCP, Principal Investigator — University of Glasgow; Salvatore Mangiafico, M.D., Ph., Principal Investigator — Careggi University Hospital; Lawrence Wong, M.D., Ph.D., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Ahmed N, Lees KR, von Kummer R, Holmin S, Escudero-Martinez I, Bottai M, Jansen O, Wahlgren N; Collaborators. The SITS Open Study: A Prospective, Open Label Blinded Evaluation Study of Thrombectomy in Clinical Practice. Stroke. 2021 Mar;52(3):792-801. doi: 10.1161/STROKEAHA.120.031031. Epub 2021 Feb 10. PMID 33563015